CLINICAL TRIAL: NCT07213570
Title: Regorafenib as Second-line Treatment of Patients With RAS-mutant Advanced Colorectal Cancer: a Multicentre, Phase 2 Study
Brief Title: STREAM-2: Second-line Treatment With REgorafenib in Advanced RAS-Mutant Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STREAM-2; 2024-519669-23-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-22; First posted 2025-10-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer Metastatic
Keywords: metastatic colorectal cancer; liquid biopsy; Regorafenib; RAS-mutation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regorafenib for ARM A - experimental arm (Experimental): Regorafenib will be administered following a dose-escalation strategy: starting dose 80 mg/day orally with weekly escalation, per 40 mg increment up to 160 mg/day regorafenib); if no significant drug-related adverse events occurred for 21 days of a 28-day cycle. The following cycle will be administered at highest tolerated dose from cycle 1 (up to 160 mg), as per current guidelines and clinical practice.
  Treatment will continue until disease progression, unacceptable toxic effects, motivated decision to stop the treatment by the treating physician, or refusal or withdrawal of consent by the patient.
  Interventions: Drug: Regorafenib (BAY73-4506)
- Standard treatment for ARM B - calibration arm (Active Comparator): Patients will continue to receive study treatment until treatment failure as previous defined, unacceptable toxicity, physician's decision, patient's refusal, or any other discontinuation criteria.
  Interventions: Drug: standard second line treatment, at discretion of the investigator

INTERVENTIONS:
Drug: standard second line treatment, at discretion of the investigator — Combination treatment may include: 5FU/LFA, capecitabine, oxaliplatin, irinotecan, bevacizumab, aflibercept
  Arms: Standard treatment for ARM B - calibration arm
Drug: Regorafenib (BAY73-4506) — Regorafenib will be administered following a dose-escalation strategy: starting dose 80 mg/day orally with weekly escalation, per 40 mg increment up to 160 mg/day regorafenib); if no significant drug-related adverse events occurred for 21 days of a 28-day cycle. The following cycle will be administered at highest tolerated dose from cycle 1 (up to 160 mg), as per current guidelines and clinical practice.
  Treatment will continue until disease progression, unacceptable toxic effects, motivated decision to stop the treatment by the treating physician, or refusal or withdrawal of consent by the patient.
  Every cycle will be administered every 28 days (four weeks) +/- 3 days.
  Arms: Regorafenib for ARM A - experimental arm

SUMMARY:
The investigators hypothesize that patients with mCRC RAS-mutant eligible for a second line treatment with good prognostic features, identified as single metastatic site, long progression free survival (PFS) in first line treatment, might benefit from a personalized approach, with less intensive treatment with regorafenib as part of a continuum-of-care strategy aimed at ensuring quality of life and extending survival.

DETAILED DESCRIPTION:
This study is an open label, randomized, multicentric, non comparative, phase-2 study. The study population will include patients with metastatic colorectal cancer (mCRC) RAS-mutant, upon progression to first line treatment, candidate to a second line, with favourable prognostic features, defined as progression free survival >6 months in first line and/or one metastatic site at study entry. A total of 60 patients (30/arm) will be require. At the time of enrollment, patients will be randomized electronically 1:1 to one of the two arms: ARM A (experimental treatment: regorafenib) and ARM B (calibration arm: standard second line treatment, at discretion of the investigator) Each cycle will be administered every four weeks for arm A (experimental treatment: regorafenib) with a dose-escalation strategy (experimental arm) and every two weeks for arm B (calibration arm: standard second line treatment, at discretion of the investigator). Patients will continue to receive study treatment until treatment failure as previous defined, unacceptable toxicity, physician's decision, patient's refusal, or any other discontinuation criteria. All subjects who finish treatment, whichever the reason, will enter in the follow-up. All patients will be followed until death and data on subsequent treatment will be collected. All measurable and non-measurable lesions must be documented at screening (within 28 days prior to randomization) and re-assessed at each subsequent tumor evaluation (every 8 weeks). Tumor assessment by CT scan (chest, abdomen and pelvis) or MRI (abdomen and pelvis); CEA, CA 19.9; and any other tests resulted positive during baseline staging, will be performed at week 8 and every 8 weeks during treatment until treatment failure in both arms. Patients discontinuing study treatment without progressive disease, will undergo tumor assessments every 8 weeks until progressive disease or study withdrawal. Toxicities will be evaluated at each clinical visit throughout the study treatment and up to 4 weeks after last cycle of treatment accordingly to the Common Terminology Criteria for Adverse Events (AEs) of the National Cancer Institute (CTCAE-NCI) version 5.0. Quality of Life will be assessed by the EORTC QLQ-C30 v.3.0 and QLQ-CR29 questionnaire that will be completed by patients at baseline (prior to treatment, once eligibility is confirmed) and every 8 weeks until disease progression, treatment failure or death. At the same time points will be administered selected items of PRO (Patients Reported Outcome) -CTCAE questionnaire and financial toxicity assessed through the PROFFIT questionnaire. Blood samples will be collected at baseline, during treatment, and at progression. Biomarkers will be correlated with clinical response, patient outcome and toxicity. In addition, biomarkers will be evaluated on tumor tissues from primary tumors or metastases at baseline, when available.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to study procedures and to correlative studies.
2. Either sex aged ≥ 18.
3. Histologically proven of colorectal adenocarcinoma.
4. Diagnosis of metastatic disease.
5. RAS mutant at initial diagnosis assessed at local centers according with a validated method defined by EMA and known MMR/MSI status.
6. Achieved a PFS in first line > 6 months with chemotherapy in combination to antiangiogenic treatment OR with one metastatic site at study entry
7. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1 at study entry.
8. Imaging-documented measurable disease, according to RECIST 1.1 criteria.
9. Estimated life expectancy of more than 12 weeks
10. Adequate bone marrow hematological function: absolute neutrophil count (ANC) ≥ 1.5 x 109/L and platelet count ≥ 100 x 109/L and hemoglobin ≥ 9 g/dL.
11. Adequate liver function: total bilirubin ≤ 1.5 x upper limit of normal (ULN) or ≤ 2 (in case of biliary stent) and aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 5 X ULN.
12. Adequate renal function: serum creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min in males and ≥50 mL/min in females (calculated according to Cockroft-Gault formula).
13. Electrolytes (i.e. magnesium, calcium, sodium and potassium) within laboratory normal range.
14. Known dihydropyrimidine dehydrogenase (DPYD) activity is mandatory. Additional analysis of polymorphisms uridine diphosphate-glycosyltransferase 1 (UGT1A1) enzyme is recommended but not mandatory.

Exclusion Criteria:

1. Prior malignancy within five years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
2. Any contraindication to regorafenib.
3. Not received immunotherapy if dMMR or MSI-H.
4. Major surgical intervention within 4 weeks prior to enrollment.
5. Pregnancy and breast-feeding.
6. Any brain metastasis.
7. Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study, or which would jeopardize compliance with the protocol, or would interfere with the results of the study.
8. History of poor co-operation, non-compliance with medical treatment, unreliability or any condition that may impair the patient's understanding of the Informed consent form.
9. Participation in any interventional drug or medical device study within 30 days prior to treatment start.
10. Sexually active males and females (of childbearing potential) unwilling to practice contraception (barrier contraceptive measure or oral contraception) during the study and until 6 months after the last trial treatment.
11. Complete deficiency of activity of dihydropyrimidine dehydrogenase (DPYD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival rate at 6 months in the two arms. | up to 6 months from randomization
  Progression Free Survival rate at 6 months(PFS rate at 6-months) is defined as the rate of assessable patients alive and not progressed after 6 months from study initiation (i.e randomization) to the first documentation of objective disease progression by RECIST 1.1 criteria, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression free survival (PFS) | up to 1 year last patients randomized
  Progression free survival (PFS) calculated as the time from randomization until the date of death from any cause until the date of the first observation of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | up to 1 year last patients randomized
  Overall survival (OS) calculated as the time from randomization until the date of death from any cause.
Objective Tumor Response Rate (ORR) | up to 1 year last patients randomized
  Objective Tumor Response Rate (ORR) assessed according to RECIST criteria 1.1, as the proportion of patients achieving complete or partial response relative to total enrolled patients.
Disease Control Rate (DCR) | up to 1 year last patients randomized
  Disease Control Rate (DCR) defined as the proportion of patients with complete/partial response and stable disease as their best response
Progression free survival 2 (PFS2) | up to 1 year last patients randomized
  Progression free survival 2 (PFS2) calculated as the time from registration to progression from subsequent line of treatment or death without progression, whichever occurred first.
Overall Toxicity rate | up to 1 year last patients randomized
  Overall Toxicity rate defined as adverse events graded according NCI CTCAE v 5.0. as the proportion of patients experiencing any grade AE accordingly to the NCI Common Terminology Criteria of Adverse Events (NCI CTC-AE) Version 5, relative to the total of patients receiving at least one cycle of treatment.AE will be listed individually by the patient and summarized overall (severity grades 1-4) and for grade ≥3 by treatment received.
Quality of life (QoL) | questionnaires must be completed before any study procedure but within 2 weeks prior to randomization (baseline) and thereafter every 8 weeks from randomization until disease progression, treatment failure or death, assessed up to 18 months
  Quality of life (QoL) investigated through the EORTC QOL-C30 questionnaires at baseline (prior to treatment start, once eligibility is confirmed) and every 8 weeks from randomization until disease progression, treatment failure or death.
Quality of life (QoL) | questionnaires must be completed before any study procedure but within 2 weeks prior to randomization (baseline) and thereafter every 8 weeks from randomization until disease progression, treatment failure or death, assessed up to 18 months.
  Quality of life (QoL) investigated through the EORTC QOL-CR29 questionnaires at baseline (prior to treatment start, once eligibility is confirmed) and every 8 weeks from randomization until disease progression, treatment failure or death.
PRO-CTCAE | questionnaires must be completed before any study procedure but within 2 weeks prior to randomization (baseline) and thereafter every 8 weeks from randomization until disease progression, treatment failure or death, assessed up to 18 months.
  PRO-CTCAE questionnaires will be administered at the same time points with items dedicated in particular to Hand-Foot Syndrome and Hand-Foot skin reactions, diarrhea and neuropathy, to better evaluate the effect of two different strategies of treatment on the health-related QoL.
Financial toxicity assessed through the PROFFIT questionnaire | at baseline (prior to treatment start, once eligibility is confirmed) and every 8 weeks from randomization until disease progression, treatment failure or death, assessed up to 18 months.
  Financial toxicity assessed through the PROFFIT questionnaire at baseline (prior to treatment start, once eligibility is confirmed) and every 8 weeks from randomization until disease progression, treatment failure or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Nazionale Tumori | "Fondazione Pascale", Napoli, Italy, Italy